CLINICAL TRIAL: NCT04685512
Title: Effect of Tenofovir/Emtricitabine Short Course on Viral Clearance in Patients Recently Infected With SARS-COV2 (Covid-19) Not Requiring Hospitalization: a Phase IIB/III Multicenter Open-label Randomized Controlled Trial
Brief Title: Effect of Tenofovir/Emtricitabine in Patients Recently Infected With SARS-COV2 (Covid-19) Discharged Home
Acronym: AR0-CORONA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-070
Record Dates: First submitted 2020-11-16; First posted 2020-12-28 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; TDF/FTC; ambulatory patients; Replication rate of the virus
MeSH Terms: conditions — COVID-19 | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Phase 2B: 30 treated, 30 untreated - 1 interim analysis planned after inclusion of 30 patients / Phase 3: 90 treated, 90 untreated - 2 interim analyses planned after inclusion of 60 and 120 patients
Who Masked: Outcomes Assessor
Masking Description: Biologists in Endpoint Adjudication committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDF / FTC (Experimental): 2 tablets on Day-1 then 1 tablet/day for 6 days
  Interventions: Drug: tenofovir disoproxil and emtricitabine
- usual care (No Intervention): Standard of Care

INTERVENTIONS:
Drug: tenofovir disoproxil and emtricitabine — Experimental drugs administration of 7-day short course TDF/FTC
  Arms: TDF / FTC

SUMMARY:
COVID-19 pandemic is currently affecting the globe. To date, there is no effective oral therapy against SARS-CoV2 infection. The investigators propose to test as a repurposing drug combination, a short course of tenofovir disoproxil and emtricitabine (TDF/FTC), as a proof-of-concept randomized open-label study to test its viral efficacy against SARS-CoV2.

DETAILED DESCRIPTION:
The SARS-CoV2 pandemic is causing morbidity and mortality. There is no cure. Remdesivir is a nucleotide analogue that has demonstrated its efficacy in vitro against SARS-CoV2 and in humans (shorten symptoms duration by 2 days without improving survival), but it is used parenterally. TDF belongs to the same therapeutic class, represents a promising avenue of research. TDF/FTC demonstrated in vivo efficacy against SARS-CoV2 in preclinical animal models and its use is associated with reduced risk of SARS-CoV2 infection in 2 large cohorts of HIV infected patients.The objective of this work is to evaluate the anti-viral efficacy of the TDF/FTC combination in short course in patients infected with SARS-CoV2 on an outpatient basis.

The investigators propose a multicenter, open-label, phase 2B/3 randomized trial of a 7-day treatment with TDF / FTC (2 tablets on Day-1 then 1 tablet / day for 6 days) according to the dosage used in pre-exposure prophylaxis for HIV. This study should include 60 outpatients (Phase 2B) and 120 additional outpatients (Phase III) who were diagnosed with SARS-CoV2 positive and with no contraindication to TDF / FTC and without criteria for hospitalization. The primary endpoint of the phase 2B will be the SARS-CoV2 antiviral efficacy quantified by RT-PCR nasopharyngeal sample Ct increase on Day-4 compared to baseline. The primary endpoint of the phase 3 will be the rate of non-contagious PCR on Day-4 from a nasopharyngeal sample. Secondary endpoints will be tolerance, symptoms resolution, percentage of hospitalization and the rate of non-contagious PCR on Day-7 from a nasopharyngeal sample.

The investigators hypothesize that compared to no treatment, treatment with TDF/FTC reduces at Day-4:

* SARS-CoV2 viral load corresponding to a 4-point +/-5 increase in Ct (Phase 2B)
* contagious carriage from 80% to 60% (Phase 3).

The AR0-CORONA investigators hope, through this study, to be able to validate an anti-viral treatment making it possible to reduce the duration of contagiousness and thus contribute to attenuating the R0 of recently infected patients carrying SARS-CoV2 who are isolated at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and over
* SARS-CoV2 Infection confirmed by PCR
* Patients who do not require immediate hospitalization
* Signed informed consent

Non-Inclusion criteria:

* Patients with HIV or Hepatitis B
* Symptoms suggestive of a SARS-CoV2 infection that has been progressing for more than 7 days
* Asympomatic patients with unknown date of infection or date of infection>7 days
* Chronic HCV infection
* Contraindication to the use of TDF/FTC
* Hypersensitivity to tenofovir, to emtricitabine or to any of the excipients (especially lactose)
* Glomerular filtration rate <80mL / min
* Recent (less than 7 days) or concomitant use of NSAIDs or other nephrotoxic drugs (antiinfectives, immunosuppressants, allopurinol, lithium
* need for hospitalization for contemporary decompensation of a comorbidity
* need for hospitalization due to SARS-CoV2 infection:
* Capillary oximetry less than 95%
* clinical evaluation by the investigating doctor leading to hospitalization
* Pregnant or breastfeeding women

Exclusion Criteria:

- Diagnosis of pregnancy during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Phase 2B: Reduction of SARS-CoV2 viral load assessed by Ct PCR at day-4 adjusted on Ct PCR SARS-CoV2 viral load at baseline (ANCOVA) | Day-4 after the start of study
  Nasopharyngeal swab performed at baseline and day-4 with RT-PCR for SARS-CoV2
Phase 3: Rate of non-contagious nasopharyngeal sample for SARS-CoV2 by PCR on Day-4 with Ct > or = 28 | Day-4 after the start of study
  Nasopharyngeal swab performed at day-4 with RT-PCR for SARS-CoV2

SECONDARY OUTCOMES:
Phase 2B/3: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the start of the study to Day-7
  Number of adverse events according to the CTCAE grade
Phase 3: Symptoms score | From the start of the study to Day-7
  Self-reported COVID-19 related symptoms
Phase 3: Proportion of secondary hospitalization | Day-15
  Assessed by investigators up to day-15
Phase 3: Rate of non-contagious nasopharyngeal sample for SARS-CoV2 by PCR on Day-7 with Ct > or = 28 | Day-7 after the start of study
  Nasopharyngeal swab performed at day-7 with RT-PCR for SARS-CoV2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Parienti, Principal Investigator — University Hospital, Caen
Locations (2):
- France (2):
  - Caen University Hospital, Caen, Calvados
  - Regional Hospital, Orléans

IPD SHARING:
Plan to Share IPD: Yes
We encourage contact the corresponding author for academic IPD sharing

REFERENCES:
- [Result] Parienti JJ et al. EClinicalMedicine 2021: https://authors.elsevier.com/sd/article/S2589-5370(21)00273-X
- [Derived] Parienti JJ, Prazuck T, Peyro-Saint-Paul L, Fournier A, Valentin C, Brucato S, Verdon R, Seve A, Colin M, Lesne F, Guinard J, Ar Gouilh M, Dina J, Vabret A, Hocqueloux L. Effect of Tenofovir Disoproxil Fumarate and Emtricitabine on nasopharyngeal SARS-CoV-2 viral load burden amongst outpatients with COVID-19: A pilot, randomized, open-label phase 2 trial. EClinicalMedicine. 2021 Aug;38:100993. doi: 10.1016/j.eclinm.2021.100993. Epub 2021 Jun 27. PMID 34222849